CLINICAL TRIAL: NCT06567093
Title: Effect of Leg and Heel Massage on Pain Experienced During Heel Blood Collection and Physiological Parameters in Newborns: Randomized Controlled Study
Brief Title: Effect of Leg and Heel Massage on Pain During Heel Blood Collection Newborns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Aylin Kurt, Asst. Prof., Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024-SBB-0076
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Pain; Infant ALL
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): All registered participants in the intervention group, will receive the leg and heel massage before the the heel blood collection.
  Interventions: Other: Baby Foot and Leg Massage
- Control (No Intervention): All registered participants in the intervention group, will receive the routine care before the leg and heel massage before the the heel blood collection.

INTERVENTIONS:
Other: Baby Foot and Leg Massage — Baby Foot Massage stages
  * The baby is placed on his back, either on the bed or on the couch.
  * One of the baby's feet is lifted into the air by grasping the back of the ankle.
  * Start stroking with circular movements, starting from the heel and moving up to the toes. Stroking should be done with the thumb.
  * Here, it might be good to get between the toes.
  * The same procedure is applied to the other foot.
  * Massage is continued until it is noticed that the baby calms down.
  Baby Leg Massage stages
  * Start by lifting the leg to be massaged.
  * Here, the palms of both hands are used. The baby's leg is placed between both hands and the leg is stroked by moving the palms in opposite directions. This movement is continued from above the ankle to the hip.
  * The same procedure is applied to the other leg.
  * Massage is continued until the baby calms down.
  Arms: Experimental

SUMMARY:
This study was planned to evaluate the effect of leg and heel massage on newborns, the pain experienced during heel blood collection, and the effects on physiological parameters.

H1: Newborn Infants Pain Scale scores are lower in leg and heel massage group than control group.

H2: Heart rates are lower in leg and heel massage group than control group. H3: Oxygen saturation levels are higher in leg and heel massage group than control group.

DETAILED DESCRIPTION:
In this study, there will be two groups as the intervention (who will receive leg and heel massage) and the control group (who will receive routine care). A power analysis was performed based on the number of children in both groups, based on another study using the scales to be used in the research. According to the calculations made in the G-Power 3.1 Demo package program, when the effect size was accepted as 0.8, it was seen that at least 30 cases in each group would be sufficient for 80% power. Infants who meet the research criteria will be randomly assigned to the intervention and control groups via http://www.randomize.org/ by assigning a number to the order of arrival at the hospital. The heel blood collection will be applied to both the intervention and control groups. For children in the massage group, the massage will be applied to both legs and heels of the baby. Immediately before the procedure, each leg and heel will be massaged for three minutes. The control group will receive heel blood collection with routine care. A researcher and a nurse were employed for the heel blood collection both for the intervention and control groups. A pediatric nurse performed the heel blood collection for all infants and the other researcher helped the children to assess their pain, heart rates and Oxygen saturation. Measurements 5 minutes before the heel prick procedure, during the procedure (1st minute) and 5 minutes after the heel prick application. The heel blood collection will be performed by the same nurse both in the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age is 38-41 weeks,
* The birth weight of the newborn is >2500 g
* Vital signs should be stable before the procedure,
* Postanatal age is between 2-28 days,
* There are no contraindications for the application of massage
* Delivery of the newborn to the mother after birth
* Permission of the parents of the newborn participating in the research
* Fasting period less than 3 hours/fed 30 minutes before
* A newborn who does not cry before heel blood is taken

Exclusion Criteria:

* Newborns who need respiratory support,
* Newborns with any neurological disorders (seizures)
* Newborns using opioids or babies born to mothers using opioids
* Newborns taking muscle relaxants, sedatives, analgesics
* Babies with major congenital anomalies
* Babies with an APGAR score of less than 7 in 5 minutes,
* Newborns who have undergone any surgery
* Newborns with birth trauma (especially rapid births)
* There are situations that may prevent communication with parents (e.g. language problems).
* problem)
* Newborns planned to be transferred to another hospital

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Difference of the mean score of the "Newborn Infants Pain Scale" between intervention and control groups | 9 months
  Pain assessment will be made with the "Newborn Infants Pain Scale". The "Newborn Infants Pain Scale" will be measured again during the heel prick procedure (at the 1st minute) and 5 minutes after the heel prick. At the end of the study, the change of the mean score of "Newborn Infants Pain Scale" between intervention and control groups will be examined. Data will be analyzed using Statistical Package for the Social Sciences package program.

SECONDARY OUTCOMES:
Difference of the mean score of the heart rate peak between intervention and control groups | 9 months
  Heart rate peak, which is a physiological parameter, will be evaluated. During the heel prick procedure (at the 1st minute) and 5 minutes after the heel prick application, the heart rate will be measured again. At the end of the study, the change of the mean score of "peak heart rate" between intervention and control groups will be examined. Data will be analyzed using Statistical Package for the Social Sciences package program.
Difference of the mean score of the oxygen saturation between intervention and control groups | 9 months
  Oxygen saturation value, which is a physiological parameter, will be evaluated. Oxygen saturation will be measured again during the heel prick procedure (at the 1st minute) and 5 minutes after the heel prick application. At the end of the study, the change of the mean score of "oxygen saturation" between intervention and control groups will be examined. Data will be analyzed using Statistical Package for the Social Sciences package program.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months